CLINICAL TRIAL: NCT02268760
Title: Safety, Tolerance, and Pharmacokinetics of Single Oral Doses of 5 mg, 20 mg, 60 mg, 100 mg, 200 mg, 400 mg, 600 mg, 800 mg, 1000 mg, 1200 mg, 1500 mg, 2000 mg and 2400 mg BILN 2061 ZW (PEG 400: Ethanol Solution) in Healthy Male Subjects, Combined With Preliminary Evaluation of Food Effect of the Dose of 200 mg (Two-Stage Trial Design With Randomised Double Blind Placebo Controlled Rising Dose Part and Subsequent Open Intraindividual Comparison Part)
Brief Title: Safety, Tolerance, and Pharmacokinetics of BILN 2061 ZW in Healthy Male Subjects, Combined With Preliminary Evaluation of Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 605.1
Record Dates: First submitted 2014-10-17; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — BILN 2061

ARMS (4):
- BILN 2061 ZW single rising doses (Experimental)
  Interventions: Drug: BILN 2061 ZW single rising doses
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BILN 2061 ZW fixed dose fed (Experimental)
  Interventions: Drug: BILN 2061 ZW fixed dose; Other: Standardized breakfast
- BILN 2061 ZW fixed dose fasted (Active Comparator)
  Interventions: Drug: BILN 2061 ZW fixed dose

INTERVENTIONS:
Drug: BILN 2061 ZW single rising doses
  Arms: BILN 2061 ZW single rising doses
Drug: Placebo
  Arms: Placebo
Drug: BILN 2061 ZW fixed dose
  Arms: BILN 2061 ZW fixed dose fasted; BILN 2061 ZW fixed dose fed
Other: Standardized breakfast
  Arms: BILN 2061 ZW fixed dose fed

SUMMARY:
To assess the safety, tolerance and pharmacokinetics of 5 mg to 2400 mg BILN 2061 ZW

1. In rising single doses
2. With and without a 64 g fat breakfast at one selected dose

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age ≥ 18 and ≤ 50 years
* Broca ≥ - 20 % and ≤ + 20 %

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders, including a history of viral hepatitis, or serological evidence of active Hepatitis B or Hepatitis C infection
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 1 month prior to administration or during the trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range and of clinical relevance
* History of any familial bleeding disorder

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2001-06; Primary Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically relevant changes in vital signs (systolic and diastolic blood pressure, pulse rate) | Pre-dose, up to 48 hours after drug administration
Changes from baseline in laboratory tests | Pre-dose and 48 hours after drug administration
Number of patients with clinically relevant changes in 12-lead ECG | Pre-dose, up to 48 hours after drug administration
Changes from baseline in physical examination | Pre-dose and 48 hours after drug administration
Number of patients with adverse events | Up to 48 hours after drug administration
Global assessment of tolerability by the investigator on a 4-point scale | Up to 48 hours after drug administration
Maximum concentration of the analyte in plasma after a single dose administration (Cmax) | up to 48 hours after drug administration
Area under the concentration-time curve of the analyte in plasma from time 0 to infinity (AUC0-infinity) | up to 48 hours after drug administration
Time to reach Cmax following a single dose administration (tmax) | up to 48 hours after drug administration
Elimination half-life of the analyte in plasma (t1/2) | up to 48 hours after drug administration
Total oral clearance of the analyte from plasma after oral administration, divided by F (bioavailability factor) (CL/F) | up to 48 hours after drug administration
Total mean residence time of the analyte in plasma (MRT) | up to 48 hours after drug administration
Apparent volume of distribution during the terminal elimination phase (Vz/F) | up to 48 hours after drug administration
Amount of intact drug excreted in urine (Au) | up to 48 hours after drug administration